CLINICAL TRIAL: NCT06707857
Title: Effects of Tendon Neuroplastic Training on Pain, Range of Motion and Disability in Patients With Rotator Cuff Tendinopathy
Brief Title: Effects of TNT on Pain, ROM and Disability in Patients With RC Tendinopathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0111
Record Dates: First submitted 2024-11-25; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Rotator Cuff Tendinopathy
Keywords: Rotator cuff tendiopathy; Tendon neuroplastic training; Disability; Range of motion; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: In this parallel- group randomized control trial(RCT) Rotator cuff tendinopathy patients will be assigned to either tendon neuroplastic training or to traditional treatment plan. this study aims to evaluate the effects pf tendon neuroplastic training on pain, range of motion and disability.
Who Masked: Outcomes Assessor
Masking Description: The study was single blinded, as accessor of the study were kept blind to the intervention groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tendon neuroplastic training (Experimental): Group A will be treated with tendon neuroplastic training. The exercise involved isolated abduction external rotation ,internal rotation and flexion paced to an external audio cue on the patients' smartphone The patient was to listen to the sound and track the movement of the metronome with his eyes, as pacing to these types of external cues has been shown to modulate conspiratorial excitability.The pace of the metronome was set to 6 beats per minute such that each beat was ten seconds apart. This allowed a ten second isometric, eccentric and concentric phase, in 30 seconds totally. Three sets of 10 repetitions of slow progressive exercises (eccentric, concentric and isometric respectively) of the wrist rotator cuff muscles at each treatment session were performed, with 1-min rest interval between each set.
  The patient followed the supervised exercise programme 3 times a week for 6 weeks
  Interventions: Other: tendon neuroplastic training
- Conventional training (Active Comparator): Group B will be treated with conventional therapy Participants will perform isometric contraction of the arm at 90° of elevation in the scapular plane. External and internal rotation, respectively) will be performed in the same positions of isometric strength assessment.Individuals will perform three sets, sustained for 32 s, at 70% of maximal voluntary isometric contraction (MVIC), resting for 80 seconds between sets.Resistance load will be determined according to maximal isometric strength of elevation and external and internal rotations measured during the pre-intervention assessment
  Interventions: Other: conventional training

INTERVENTIONS:
Other: tendon neuroplastic training — Throughout the training, participants pain, range of motion and disability were monitored and they were asked to report any discomfort or unusual sign.
  Arms: Tendon neuroplastic training
Other: conventional training — Throughout the training, participants pain, range of motion and disability were monitored and they were asked to report any discomfort or unusual sign.
  Arms: Conventional training

SUMMARY:
EFFECTS OF TENDON NEUROPLASTIC TRAINING ON PAIN, RANGE OF MOTION AND DISABILITY IN PATIENTS WITH ROTATOR CUFF TENDINOPATHY

DETAILED DESCRIPTION:
Rotator cuff tendinopathy is a condition where the shoulder's tendon suffers small tears or inflammation, often causing pain frequently arises from repetitive overuse or the natural aging process Regular overhead activities can aggravate the shoulder's wear and tear, leading to tendinosis. The purpose of this study is to evaluate and compare the impact of tendon neuroplastic training with standard treatments on pain levels, functional disability, and the range of motion in patients suffering from rotator cuff tendinopathy. Data were collected from Riphah rehabilitation clinic Lahore. Nprs , goinmeter and Spadi questioner were used before and after the intervention. Assessment was done through the tool before and after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Have a current shoulder complaint lasting at least three months prior to the time of enrollment
* Pain is located in the proximal lateral aspect of the upper arm (C5 dermatome)
* Positive Hawkins-Kennedy test

Exclusion Criteria:

* Bilateral shoulder pain
* Less than 90 degrees of active elevation of the arm
* Corticosteroid injection within the last six weeks
* Radiologically verified fracture
* Glenohumeral osteoarthritis
* Surgery or dislocation of the affected shoulder
* Symptomatic arthritis in the Ac joint
* Frozen shoulder
* Symptoms derived from the cervical spine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Numeric pain rate scale (NPRS) | 6 weeks
  Patient level of pain will be assessed using this scale. This scale ranges from 0 to 10. 0 indicates "no pain" and 10 indicates "worst pain".
Shoulder pain and disability index (spadi) | 6 weeks
  Patient level of disability will be assessed using this scale. This ranges from 0 to 100. 0 indicates no disability" and 100 indicates disability"
Universal Goniometer (UG) | 6 weeks
  It will measure range of motion of shoulder

CONTACTS AND LOCATIONS:
Overall Officials: Saba Rafique, MS-OMPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah Rehabilitation clinic, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No